CLINICAL TRIAL: NCT00731354
Title: A Multi-Center, Prospective, Randomized, Single-Blind, Controlled Clinical Trial Comparing VASER-Assisted Lipoplasty and Suction-Assisted Lipoplasty.
Brief Title: VASER-Assisted Lipoplasty Compared With Suction-Assisted Lipoplasty
Acronym: Contra-Lateral
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sound Surgical Technologies, LLC. (Industry)
Responsible Party: Amber Eruchalu, M.S., CCRP./ Clinical Program Manager, Sound Surgical Technologies, LLC
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: SST40.2
Record Dates: First submitted 2008-08-04; First posted 2008-08-11 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Healthy
Keywords: lipoplasty; liposuction; VASER; body contouring; body sculpting; Any patient; expressing; interest; in elective surgery
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAL (Active Comparator): Each patient will have Suction Assisted Lipoplasty procedure on one side of the body (this will be considered the control side)
  Interventions: Device: Suction-assisted Lipoplasty
- VAL (Active Comparator): Each patient will have VASER- assisted lipoplasty on the opposite side of the body. This will be the comparison side.
  Interventions: Device: VASER-assisted lipoplasty

INTERVENTIONS:
Device: Suction-assisted Lipoplasty — Standard Suction-assisted lipoplasty will be performed on one side of the body to remove excess fat and contour the body in one or more of the following body areas: arm, inner thigh, outer thigh, back
  Other Names: Suction-assisted lipoplasty, Liposuction
  Arms: SAL
Device: VASER-assisted lipoplasty — VASER-assisted lipoplasty will be performed on the opposite side of the body to remove excess fat and contour the body in one or more of the following body areas: arm, inner thigh, outer thigh, back
  Other Names: VAL, VASER, LipoSelection, 3rd Generation UAL
  Arms: VAL

SUMMARY:
This study is being done to compare two commonly available types of body contouring, VASER-Assisted Lipoplasty (VAL) and Suction-Assisted Lipoplasty (SAL), and to decide if one procedure is preferred by patients and/or surgeons over the other. Participants will have VAL on one side of their body and SAL on the opposite side.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary, signed informed consent in accordance with institutional policies
* be between the ages of 18-50 years old
* Be willing and able to appear for all scheduled, post-operative visits with their doctor
* Have moderate to good skin tone
* Have excess fatty tissue in the arms, medial thighs, lateral thighs, or back where the extra tissue is expected to be composed of adipose tissue.
* Have a body mass index between 20-30
* Are non-smokers

Exclusion Criteria:

* under the age of 18
* over the age of 50
* are undergoing boy contouring for reconstruction following injury or disease are deemed inappropriate candidates for surgery due to medical or mental health reasons
* are concurrently being treated with other investigational agents or have participated in an investigational study within 60 days prior to surgery
* elect not to participate in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Investigators aim to assess outcomes associated with the two different methods to determine if one technology/technique offers superior results compared to the other. | 6 months

SECONDARY OUTCOMES:
To assess the difference in patients' post-operative pain level between the SAL side and the VAL side | 6 months
To assess the difference in patients' post-operative sensation level between the SAL side and the VAL side | 6 months
To assess the difference in post-operative patient preference between the SAL side and the VAL side | 6 months
To assess the difference in post-operative ecchymosis between the SAL side and the VAL side | 6 months
To assess the difference in post-operative skin retraction between the SAL side and the VAL side | 6 months
To assess the difference in the amount of aspirate blood content between the SAL side and the VAL side | 1 day
To assess any difference in the amount or degree of complications using the the SAL procedure versus the VAL procedure | 6 months
To assess the difference in the time required for the SAL procedure versus the time required for the VAL procedure. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Onelio Garcia, MD, F.A.C.S, Principal Investigator — Plastic Surgery Center of South Florida; Michael Nagy, MD, F.A.C.S, Principal Investigator — Personal Enhancement Center; Paul F Vanek, MD, F.A.C.S., Principal Investigator — Lake Hospital Systems
Locations (3):
- United States (3):
  - Plastic Surgery Center of South Florida, Miami, Florida
  - Personal Enhancement Center, Toms River, New Jersey
  - Paul F. Vanek, M.D., F.A.C.S., Mentor, Ohio

REFERENCES:
- See also: Sound Surgical Technology - technique description — http://www.vaser.com/